CLINICAL TRIAL: NCT06005389
Title: Serum Galectin-3: A Potential Marker of Human Papillomavirus Infection Before and After Treatment of Cutaneous Warts
Brief Title: Serum Galectin-3 as a Marker of Human Papillomavirus Infection
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Hasan Sayed, lecturer, Assiut University
Other Study IDs: Galectin-3 and HPV infection
Record Dates: First submitted 2023-08-04; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Human Papillomavirus Infection
Keywords: Galectin-3; Human papillomavirus; Warts; Cryotherapy
MeSH Terms: conditions — Papillomavirus Infections; Warts | interventions — Cryotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 50 patients with common or planter cutaneous warts: Every patient had a cryotherapy session every 2 weeks until complete clearance for a maximum of six sessions and follow-up was done at 3 months after treatment completion to detect any recurrence. The therapeutic efficacy was evaluated by a decrease in the size (measured by a ruler) and the number of warts with photographic documentation at (the baseline, each visit, 2 weeks after the final session, and the 3 months follow-up period). The response of the treated wart was considered: complete; if there was a disappearance of the wart and appearance of normal skin markings, partial; if the warts had regressed in size or decreased in number and no response; if no decrease in wart size or number.
  From each patient 3 ml venous blood was withdrawn under complete aseptic conditions before treatment and 2 weeks after the last treatment session by a disposable plastic syringe. Serum Gal-3 was measured using human Galectin-3 enzyme-linked immunosorbent assay (ELISA) kits.
  Interventions: Procedure: cryotherapy; Diagnostic Test: serum Galectin-3 assay
- 50 healthy age-and sex-matched control subjects.: From each control subject, 3 ml venous blood was withdrawn under complete aseptic conditions before treatment and 2 weeks after the last treatment session by a disposable plastic syringe. Serum Gal-3 was measured using human Galectin-3 enzyme-linked immunosorbent assay (ELISA) kits.
  Interventions: Diagnostic Test: serum Galectin-3 assay

INTERVENTIONS:
Procedure: cryotherapy — Every patient had a cryotherapy session every 2 weeks until complete clearance for a maximum of six sessions and follow-up was done at 3 months after treatment completion to detect any recurrence. Each wart was frozen using the spray technique by CRY-AC Liquid Nitrogen Dispenser Brymill, USA for 10 to 30 seconds until a 1- to 2-mm ice ball halo was formed surrounding the targeted area.
  Groups: 50 patients with common or planter cutaneous warts
Diagnostic Test: serum Galectin-3 assay — From each patient and control, 3 ml venous blood was withdrawn under complete aseptic conditions before treatment and 2 weeks after the last treatment session by a disposable plastic syringe; the collected blood was placed on a plain tube without anticoagulant for 30 min at room temperature till coagulation occurs; after this, centrifugation of tubes was done for 20 min at 1000 rpm. The serum was separated into an aliquot and placed at -20 degrees Celsius for further analysis. Serum Gal-3 was measured using human Galectin-3 enzyme-linked immunosorbent assay (ELISA) kits supplied by ELK Biotechnology CO., LTD, Wuhan, China, catalog number (ELK2790) based on the Sandwich-ELISA technique as per the manufacturer's instructions.

SUMMARY:
This study aimed to assess the serum Galectin-3 levels in patients with warts both before and after cryotherapy and to investigate its potential contribution to the pathogenesis of human papillomavirus infection.

DETAILED DESCRIPTION:
Galectin-3 regulates many functions at the cellular level such as cell attachment, proliferation, and apoptosis. Numerous viral illnesses, including human papillomavirus infection, were reported to have elevated serum levels of Galectin-3. .

Methods: Fifty patients suffering from warts, and fifty healthy controls were included in this study. Enzyme-linked immunosorbent assay was used to measure serum levels of Galectin-3 both before and 2 weeks after the last cryotherapy session.

ELIGIBILITY:
Inclusion criteria:

1. Patients with non-genital warts.
2. Age of patients: from 18 to 60 years.

Exclusion criteria:

1. Patients with genital and mucosal warts.
2. Pregnancy and breastfeeding.
3. Patients who received any wart treatment during the last month before enrollment in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This case-control study was performed on 50 patients with any type of cutaneous warts except for genital warts and 50 apparently healthy age-and sex-matched control subjects without a history of warts attending the Outpatient Clinic of Dermatology, Venereology and Andrology Department of Assiut University Hospitals.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Serum Galectin-3 levels assessment in patients with cutaneous warts. | 1 year
  3 ml of venous blood from each patient and control was drawn under strict aseptic conditions employing a single-use plastic syringe. Once the blood had been collected, it was put in a simple tube without an anticoagulant and left there for 30 minutes at room temperature until coagulation had taken place. The tubes were then centrifuged at 1000 rpm for 20 minutes. For further examination, an aliquot of the serum was taken and stored at 20 degrees Celsius. Human Galectin-3 enzyme-linked immunosorbent assay (ELISA) kits with the catalogue number (ELK2790) from ELK Biotechnology CO., LTD, Wuhan, China, were used to quantify serum Gal-3 in accordance with the manufacturer's instructions.
look at Galectin-3 serum level conceivable contribution to the aetiology of HPV infection, and determine how cryotherapy affected serum Galectin-3 levels. | 1 year
  All patients had a thorough medical history taken, which included information on their age, sex, occupation, the number of warts, their location, size, and past treatments, as well as any previous systemic or skin conditions or drug use. A thorough examination was performed on each patient to determine the location, kind, size, and number of warts as well as to rule out any systemic or other skin conditions.
  Before and two weeks after the last cryotherapy treatment session, serum Galectin-3 was assessed. Every patient had a cryotherapy session every 2 weeks until complete clearance for a maximum of six sessions and follow-up was done at 3 months after treatment completion to detect any recurrence. Each wart was frozen using the spray technique by CRY-AC Liquid Nitrogen Dispenser Brymill, USA for 10 to 30 seconds until an ice ball halo of 1 to 2 mm diameter encircled the intended area.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Coppock JD, Mills AM, Stelow EB. Galectin-3 Expression in High-Risk HPV-Positive and Negative Head & Neck Squamous Cell Carcinomas and Regional Lymph Node Metastases. Head Neck Pathol. 2021 Mar;15(1):163-168. doi: 10.1007/s12105-020-01195-3. Epub 2020 Jun 20. PMID 32564273